CLINICAL TRIAL: NCT04631536
Title: Managing Endothelial Dysfunction in COVID-19 : A Randomized Controlled Trial at the Lebanese American University Medical Center- Rizk Hospital
Brief Title: Managing Endothelial Dysfunction in COVID-19 : A Randomized Controlled Trial at LAUMC
Acronym: MEDIC-LAUMC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lebanese American University Medical Center (Other)
Responsible Party: Principal Investigator, Kamal Matli, Cardiology Fellow, Lebanese American University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lebanese American University
Record Dates: First submitted 2020-10-28; First posted 2020-11-17 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: Endothelial dysfunction; Nicorandil; Statin; Nebivolol; L-arginine; Folic acid
MeSH Terms: conditions — COVID-19 | interventions — Atorvastatin; Arginine; Folic Acid; Nicorandil; Nebivolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endothelial Dysfunction Protocol (Experimental): Our study will evaluate the impact of the endothelial treatment protocol (atorvastatin, nicorandil, l-arginine, folic acid and nebivolol) in patients already on optimal medical therapy for the treatment of COVID0-19 virus.
  Endothelial dysfunction protocol + Standard of Care (dexamethasone, anticoagulation, vitamin c, zinc).
  1. Atorvastatin or continue home statin Atorvastatin will be provided as a 40 mg tablet to be given PO once daily. This dose was suggested because high intensity statin has been associated with a better endothelial profile (Int J Cardiol 2017 Oct 1;244:112-118.-- Eur J Clin Pharmacol 2014 Oct;70(10):1181-93)
  2. Nicorandil Nicorandil 10 mg PO BID as the recommended dose for coronary vasodilatation by the manufacturer
  3. Nebivolol Nebivolol 2.5-5 mg PO ONCE daily while keeping Heart Rate (HR) between 50-90 bpm
  4. Folic Acid Folic Acid 5 mg po once daily
  5. L-Arginine L-Arginine 1 g po TID
  Interventions: Drug: Atorvastatin + L-arginine + Folic acid + Nicorandil + Nebivolol
- Placebo (Placebo Comparator): Placebo + Standard of Care (dexamethasone, anticoagulation, vitamin c, zinc)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin + L-arginine + Folic acid + Nicorandil + Nebivolol — active Comparator: Endothelial dysfunction protocol + Standard of Care (dexamethasone, anticoagulation, vitamin c, zinc). Treatment to be continued until 14 days or discharge/death whichever occurs first. It includes: Nebivolol 5 mg PO daily, Sigmart 10 mg PO twice daily, Atorvastatin 40 mg PO daily, Folic Acid 5 mg PO daily, L-arginine 1000 mg PO 3 times daily.
  Other Names: Nicorandil; L-arginine; Folic acid; Nebivolol
  Arms: Endothelial Dysfunction Protocol
Drug: Placebo — Placebo + Standard of Care (dexamethasone, anticoagulation, vitamin c, zinc)
  Arms: Placebo

SUMMARY:
COVID-19 infection was shown to cause endothelial dysfunction .

At the level of the endothelium the pathophysiological mechanisms have been hypothesized and were divided into pro-coagulant, pro-inflammatory, anti-fibrinolytics, impaired barrier function, vasoconstrictor and pro-oxidant. So far, the pro-coagulant and pro-inflammatory pathways have been studied and as a result dexamethasone and anticoagulation became part of the standard therapies for the disease. However, so far, no RCT has been evaluated on targeting the vasoconstrictive and antioxidant pathways with an aim of revealing clinical benefit.

So, with this trial we intend to provide a regiment composed of several medications we hypothesize will act on several downstream pathways that would improve endothelial function primarily via the increase in NO production and release.

At the time of this proposal there has been no randomized trials evaluating or testing the use of cardiovascular drugs targeting endothelial dysfunction in COVID-19 patients. As previously noted there has been a call to study these drugs and their effect after a strong research regarding their theorized effectiveness. For evidence, there was a recently published meta-analysis evaluating the role of statins in COVID-19 with preliminary findings suggested a reduction in fatal or severe disease by 30% and discredited the suggestion of harm, that emphasized on the need of well-designed randomized controlled trial to confirm the role of statins in COVID-19 patients.

Our study would help determine the potential therapeutic effect of the endothelial protocol as adjunct to mainstream management. This study seeks to further our knowledge in treating COVID-19 to ultimately improve clinical outcomes and reduce complications.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) is the novel pathogen responsible coronavirus disease 2019 (COVID-19) first discovered in Wuhan, China. Since its emergence in late December 2019, many pathophysiological mechanisms have been proposed with multiple pathways that involve various organ systems . Although considered at its emergence as a respiratory infection with manifestations ranging from lower respiratory tract infection to pneumonia and advancing to acute respiratory disease syndrome (ARDS) in its final stages, recent evidence has highlighted how disseminated the virus can be affecting almost every organ be it the heart kidneys or blood vessels . Recent trends in research have focused on elucidating the cardiovascular dysfunction in COVID-19 patients Especially following studies showing that cardiovascular risk factors are among the most common presenting comorbidities and that cardiovascular complications of SARS-CoV-2 are among the most lethal . Initial research revealed that the virus makes use of the angiotensin-converting enzyme 2 (ACE-2) receptor to infiltrate host cells. With the ACE-2 receptor being a widely expressed receptor found in multiple cells lining the lung, heart, gastrointestinal tract, kidneys and endothelial cells. Another prominent mechanism of infection is immune system dysregulation manifesting as a cytokine storm and inflammatory response over-activation.

Attempts at laying out a comprehensive or unifying pathogenesis of a COVID-19 infection have singled out endothelial dysfunction as a core pathway. The endothelium in summary is monolayer lining the arteries, veins and microvasculature. The endothelium hence plays a major role in homeostasis with interactive roles in blood pressure regulation, anti-coagulation and immune protection Moreover, it is thus relevant to note that the most common comorbidities that present with COVID-19 such as hypertension, diabetes, obesity and old age are all underlined by pre-existing endothelial damage or dysfunction. As such, endothelial dysfunction and oxidative stress and their relation to the manifestation and progression of COVID-19 infections has gain significant traction in recent publications. This breakthrough exposes several causes of endothelial dysfunction which include direct lining attack, hypoxia, cytokine storm and suppressed endothelial nitric oxide synthase (eNOS) with concomitant nitric oxide deficiency. Several studies have emphasized the role of NO signaling as a major regulator of vascular tone and its antioxidant, anti-inflammatory and antithrombotic activity. For example, augmenting the production of NO and its bioavailability by nicorandil has been proposed as a potential treatment in patients with COVID 19. Nicorandil (a vasodilatory agent composed of N-[2-hydroxyethyl]-nicotinamide nitrate) used among patients with acute heart failure emergencies However, it has never been tested in patients with cardiovascular complications resulting from COVID 19 . Statins are cardioprotective in nature with recent reports showing that they can be beneficial in COVID-19 . An important mechanism via which Statins may improve endothelial function include increasing the production of NO and subsequent vasodilation effect, along with its established major anti-inflammatory and anti-oxidant properties . Nebivolol, a cardio-selective beta blocker has also shown non-adrenergic vasodilating properties via the release of NO along with antioxidative and anti-atherosclerotic activities. Furthermore, eNOS overexpression leads to an increase in NO formation only when the BH4 synthase GTP-cyclohydrolase 1 (GCH-1) is alsoup-regulated. So, Folic Acid and L-arginine will be given to supplement our patients with BH4 . We hypothesize that its administration along with the other previously mentioned agents would improve endothelial function in patients suffering from COVID 19 via a cumulative increase in the bioavailability of Nitric Oxide (NO), and thus improving patients' outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and above admitted for inpatient treatment of COVID-19 infection
* PCR-confirmed COVID-19 classified as mild, moderate or with severe disease as per the FDA.

With mild being a positive testing by standard RT-PCR assay or equivalent test and symptoms of mild illness with COVID-19 that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea. No clinical signs indicative of Moderate, Severe, or Critical Severity.

* Moderate defined as positive testing by standard RT-PCR assay or equivalent testing and symptoms of moderate illness which could include any symptom of mild illness or shortness of breath with exertion. Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥ 20 breaths per minute, saturation of oxygen (SpO2) > 93% on room air at sea level, heart rate ≥ 90 beats per minute. No clinical signs indicative of Severe or Critical Illness Severity.
* Severe symptoms could include any symptom of moderate illness or shortness of breath at rest, or respiratory distress. Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory 468 rate ≥ 30 per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air at sea level or 469 PaO2/FiO2 < 300.
* No criteria for Critical Severity.
* Eligible for or taking statin

Exclusion Criteria:

* Participant in another RCT
* Myocarditis
* Patients who are already on beta-blockers

Patients already on Nicorandil.

. Patients taking PDE5 inhibitors or Riociguat

.Shock as defined by SBP<90 for more than 30 minutes not responding to IV fluids with evidence of end organ damage.

.Severe bradycardia (<50 bpm).

.Heart block greater than first-degree (except in patients with a functioning artificial pacemaker).

.Decompensated heart failure.

.Sick sinus syndrome (unless a permanent pacemaker is in place).

.Severe hepatic impairment (Child-Pugh class C) or active liver disease.

.Unexplained persistent elevations of serum transaminases.

.Pregnancy or breastfeeding.

.Hypersensitivity to any of the medications.

* Can't take medications orally
* Patient refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-03-29 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | From date of intervention administration until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  The primary outcome was the time to recovery, defined as the first day, during the 28 days after enrollment, on which a patient met the criteria for category 1, 2, or 3 on the eight-category ordinal scale. The categories are as follows: 1, not hospitalized and no limitations of activities; 2, not hospitalized, with limitation of activities, home oxygen requirement, or both; 3, hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infection-control or other nonmedical reasons); 4, hospitalized, not requiring supplemental oxygen but requiring ongoing medical care (related to Covid-19 or to other medical conditions); 5, hospitalized, requiring any supplemental oxygen; 6, hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices; 7, hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); and 8, death

SECONDARY OUTCOMES:
Need for ICU admission or invasive mechanical ventilation | Assessment on daily basis for up to 1 month or until hospital discharge/death whichever came first
  assess the patients in need of mechanical ventilation or ICU admission
All cause mortality | assessed for up to 1 month
  All cause mortality
Occurrence of side effects | Assessment on daily basis after intervention given for up to 1 month or until hospital discharge/death whichever came first
  Occurrence of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- LAUMCRH, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu YC, Chen CS, Chan YJ. The outbreak of COVID-19: An overview. J Chin Med Assoc. 2020 Mar;83(3):217-220. doi: 10.1097/JCMA.0000000000000270. PMID 32134861
- [Background] Yuki K, Fujiogi M, Koutsogiannaki S. COVID-19 pathophysiology: A review. Clin Immunol. 2020 Jun;215:108427. doi: 10.1016/j.clim.2020.108427. Epub 2020 Apr 20. PMID 32325252
- [Background] Mason RJ. Pathogenesis of COVID-19 from a cell biology perspective. Eur Respir J. 2020 Apr 16;55(4):2000607. doi: 10.1183/13993003.00607-2020. Print 2020 Apr. PMID 32269085
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335
- [Background] Murthy S, Gomersall CD, Fowler RA. Care for Critically Ill Patients With COVID-19. JAMA. 2020 Apr 21;323(15):1499-1500. doi: 10.1001/jama.2020.3633. No abstract available. PMID 32159735
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Hu Y, Sun J, Dai Z, Deng H, Li X, Huang Q, Wu Y, Sun L, Xu Y. Prevalence and severity of corona virus disease 2019 (COVID-19): A systematic review and meta-analysis. J Clin Virol. 2020 Jun;127:104371. doi: 10.1016/j.jcv.2020.104371. Epub 2020 Apr 14. PMID 32315817
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Background] Liu PP, Blet A, Smyth D, Li H. The Science Underlying COVID-19: Implications for the Cardiovascular System. Circulation. 2020 Jul 7;142(1):68-78. doi: 10.1161/CIRCULATIONAHA.120.047549. Epub 2020 Apr 15. PMID 32293910
- [Background] Hamming I, Timens W, Bulthuis ML, Lely AT, Navis G, van Goor H. Tissue distribution of ACE2 protein, the functional receptor for SARS coronavirus. A first step in understanding SARS pathogenesis. J Pathol. 2004 Jun;203(2):631-7. doi: 10.1002/path.1570. PMID 15141377
- [Background] Jung F, Kruger-Genge A, Franke RP, Hufert F, Kupper JH. COVID-19 and the endothelium. Clin Hemorheol Microcirc. 2020;75(1):7-11. doi: 10.3233/CH-209007. PMID 32568187
- [Background] Libby P, Luscher T. COVID-19 is, in the end, an endothelial disease. Eur Heart J. 2020 Sep 1;41(32):3038-3044. doi: 10.1093/eurheartj/ehaa623. PMID 32882706
- [Background] Ashour H, Elsayed MH, Elmorsy S, Harb IA. Hypothesis: The potential therapeutic role of nicorandil in COVID-19. Clin Exp Pharmacol Physiol. 2020 Nov;47(11):1791-1797. doi: 10.1111/1440-1681.13395. Epub 2020 Sep 9. PMID 32881062
- [Background] Kunal S, Gupta K, Gupta S. Statins in COVID-19: A new ray of hope. Heart Lung. 2020 Nov-Dec;49(6):887-889. doi: 10.1016/j.hrtlng.2020.07.012. Epub 2020 Aug 11. No abstract available. PMID 32861559
- [Background] Gornik HL, Creager MA. Arginine and endothelial and vascular health. J Nutr. 2004 Oct;134(10 Suppl):2880S-2887S; discussion 2895S. doi: 10.1093/jn/134.10.2880S. PMID 15465805